CLINICAL TRIAL: NCT02158715
Title: Assessment of Validity of Depth by PocketCPR as Sites of Smartphone on Arm
Status: Completed | Type: Observational
Sponsor: Hanyang University (Other)
Responsible Party: Principal Investigator, Joonbum Park, Assistant Professor, Soon Chun Hyang University
Other Study IDs: PocketCPR
Record Dates: First submitted 2014-05-16; First posted 2014-06-09 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-08

CONDITIONS: Chest Compression With Smartphone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Smartphone positioning during Chest compression
  Interventions: Device: Site of smartphone on chest compressor' arm

INTERVENTIONS:
Device: Site of smartphone on chest compressor' arm

SUMMARY:
For Cardiopulmonary Resuscitation(CPR) education, depth of chest compression is most important teaching point. However, the tool to feedback depth of chest compression like Resusci Annie Skill Reporter(Laedal Medical AS, Norway) is very helpful but too expensive to be used widely. In these days, smartphone free application can measure depth of chest compression in real-time. This study assess the validity of depth of chest compression by smartphone application, PocketCPR, as three sites of smartphone on arm or hand.

1. grap it in hand, 2. fix it on upper arm with arm band, 3. grap it in hand with arm band

To analyze the difference between Skill Reporter manikin and PocketCPR application, the investigators will use Intraclass Correlation Coefficient(ICC) as statistical method.

ELIGIBILITY:
Inclusion Criteria:

* Chest compressor with Basic Life Support certification
* Physician, Nurse, Emergency medical technician with more than 3 years clinical experience

Exclusion Criteria:

* Person who cannot practice normal chest compression with any reason

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Basic Life Support certtification licenced by American Heart Association
  Clinical experience more than 3 years associated with CPR
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2014-04; Primary Completion 2014-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Depth of chest compression | up to 1 month
  Depth of chest compression by reporting manikin and application of i-phone. Scale : millimeter

CONTACTS AND LOCATIONS:
Locations (1):
- Hanyang medical center, Seoul, Seoul, South Korea